CLINICAL TRIAL: NCT00405249
Title: 14-Day Randomized Double-Blind Comparative Viral Kinetic Study of Elvucitabine Versus Lamivudine Once Daily to HIv-1 Subjects With M184V
Brief Title: Safety Study of Elvucitabine in HIV-1 Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ACH-443-014A
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: HIV-1; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — dexelvucitabine

INTERVENTIONS:
Drug: elvucitabine

SUMMARY:
The purpose of this 28 day study is to assess the viral kinetics and safety of elvucitabine.

DETAILED DESCRIPTION:
This is a 14 day on treat/14 day off treatment randomized, double blind viral kinetic study of elvucitabine versus lamivudine administered once daily to HIV infected subjects with a documented M184V variant.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected, clinically stable, adults
* HIVRNA 5000 -150,000, CD4 100
* Genotypically documented M184V variant
* Receiving stable ART.

Exclusion Criteria:

* Hep B
* HIV-1 genotype for 4 protease inhibitors
* HIV-1 genotype positive for 2 NNRTI mutations
* Previous therapy with system myelosuppressive potential within 3 months of study start
* Use of Epogen or Neupogen
* History of cirrhosis
* Alcohol or drug dependence
* Inability to tolerate oral medication
* Women who are pregnant or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2006-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Squires, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States